CLINICAL TRIAL: NCT04189666
Title: Rivastigmine Patch (Exelon Patch) Compared to Melatonin Patch in Prevention of Postoperative Delirium in Elderly
Brief Title: Rivastigmine Patch Compared to Melatonin Patch in Prevention of Postoperative Delirium
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rania Maher Hussien, Lecturer of Anaesthesia and intensive care, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FMASU R58/ 2019
Record Dates: First submitted 2019-11-24; First posted 2019-12-06 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium | interventions — Rivastigmine; Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group R: patients receive Rivastigmine patch (Active Comparator): receive a Rivastigmine patch (4.6 mg) 24 h before the operation to 3 days post-operative
  Interventions: Drug: Rivastigmine Transdermal System [Exelon]
- Group M: patients receive Melatonin patch (Active Comparator): receive Melatonin patch (7 mg) 24 h before the operation to 3 days post-operative
  Interventions: Drug: Melatonin

INTERVENTIONS:
Drug: Rivastigmine Transdermal System [Exelon] — compare the ability of the drug in preventing postoperative delirium
  Other Names: Exelon
  Arms: Group R: patients receive Rivastigmine patch
Drug: Melatonin — compare the ability of the drug in preventing postoperative delirium
  Other Names: melatonin patch
  Arms: Group M: patients receive Melatonin patch

SUMMARY:
180 patients will be randomly divided into two groups 90 patients each using a computer-generated program.

Group R: 90 patients will receive a Rivastigmine patch (4.6 mg) 24 h before the operation to 3 days post-operative Group M: 90 patients will receive Melatonin patch (7 mg) 24 h before the operation to 3 days post-operative Patients in the two groups will be compared regarding incidence and severity of delirium on postoperative days 1, 2 or 3 and 7

DETAILED DESCRIPTION:
180 elderly patients American Society of Anaesthesiologists physical status I-III aged 60-85 years old undergoing major orthopaedic surgery will be included in this study The day prior to the operation all patients will be examined by an anaesthesia resident ''who is blinded to the study'' for preoperative cognitive impairment using Confusion Assessment Method. Patients with delirium were excluded from the study The 180 patients will be randomly divided into two groups 90 patients each using a computer-generated program. The patches will be given to the ward nurse who is blinded to the study to be administered to the patient 24 hours preoperative, during the operation and 3 days postoperative Group R: 90 patients will receive a Rivastigmine patch (4.6 mg) 24 h before the operation to 3 days post-operative Group M: 90 patients will receive Melatonin patch (7 mg) 24 h before the operation to 3 days post-operative On the day of the operation, patients will not receive premedication. In the operating room basic monitoring in the form of NIBP, SBP (systolic blood pressure), DBP (diastolic blood pressure), SPO2 (pulse oxygen saturation), ECG (electrocardiogram), will be attached and recorded every 30 mins. Level of intraoperative sedation will be monitored using Ramsay Sedation Scale.

Patients of both groups will receive Regional anaesthesia in the form of spinal or epidural anaesthesia according to Anaesthesia and surgical team preference and according to each case. Patient will be put in the sitting position, back will be sterilized by povidone- iodine, drapes will cover the back of the patient, L4-L5 or L3-L4 level will be palpated and local anaesthetic in the form of 1 ml of 2% lidocaine will be injected subcutaneous In case of spinal anaesthesia; a spinal needle G25 will be introduced. After appearance of CSF, heavy Marcaine will be injected intrathecally.

In case of epidural anaesthesia; a Tuohy needle will be introduced, on feeling loss of resistance a catheter will be threaded upward, secured in place, a test dose of 3 ml 2% lidocaine will be injected, then 12-18 ml of 0.5% isobaric Marcaine will be injected After completing the surgery patients will be sent to the Surgical ICU for postoperative monitoring. basic monitoring in the form of (NIBP, SPO2, ECG) will be monitored continuously and any abnormality will be recorded and managed according to the ICU protocol. All patients will be examined by the same anaesthesia resident ''who is blinded to the study'' for PD using Confusion Assessment Method (CAM) and level of sedation using RSS on the first, second, third and 7th postoperative day and for those who develop PD a CAM-S score will be done to assess the severity of PD.

And patients with delirium will be followed up and managed properly by a Neurology specialist.

Patients in the two groups will be compared regarding incidence and severity of delirium on postoperative days 1, 2 or 3 and 7 The investigator's primary outcome is to compare between the two groups regarding the incidence of developing PD among the elderly patients The secondary outcome is to compare between both groups regarding the severity of PD and level of sedation

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiologists physical status I-III,
* Aged 60-85 years old,
* Undergoing major orthopaedic surgery

Exclusion Criteria:

* History of CNS disorders, such as brain injury, stroke; mental illness; dementia
* Metabolic disorders and electrolyte disturbances
* Alcohol or drug dependence
* Secondary surgery or severe infectious complications
* Severe sensory impairment causing difficulty in communication (deafness or blindness)
* Medications affecting CNS as (Antipsychotics, Anticonvulsants, Antiparkinsonian, Antidepressants)

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
compare between the two groups regarding the incidence of developing Delirium among the elderly patients | seventh postoperative day
  incidence of developing postoperative delirium by Confusion Assessment Method which consisting of four features: it indicate delirium if features 1 and 2 are present and either feature 3 or 4 is present.

SECONDARY OUTCOMES:
compare between both groups regarding level of sedation | seventh postoperative day
  level of sedation by Ramsy Sedation Score which consists of 6 points: score 1; patient is Anxious (not sedated), 6; No response to stimulus (deeply sedated)

CONTACTS AND LOCATIONS:
Overall Officials: Rania Hussien, MD, Principal Investigator — lLecturer of Anaesthesia, Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Abassia, Egypt

IPD SHARING:
Plan to Share IPD: No